CLINICAL TRIAL: NCT04614454
Title: High Frequency Impulse Therapy for Neuropathic Pain in NMOSD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Michael, Levy M.D.,Ph.D., Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020P003301
Record Dates: First submitted 2020-10-22; First posted 2020-11-04 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Neuromyelitis Optica
MeSH Terms: conditions — Neuromyelitis Optica | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to receive treatment daily for 4 consecutive weeks versus sham, followed by an open-label phase for additional 4 consecutive weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects will be randomized to either the intervention or the control group, fitted and trained to use the home TENS device to self-administer treatment for at least one hour each day. The subjects will not know to which arm they are randomized. Neither will the study coordinator or the investigator. Only a 3rd party collaborator will know the assignment scheme and this will be revealed in blocks every time 4 subjects complete the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental arm (Experimental): Devices will be programmed by our study coordinator to provide a sham signal or the experimental signal. The location of the TENS electrodes will be determined by the location of the pain with the goal of placing the unit at the top of the dermatological level corresponding to the pain. The study coordinator will assist each subject to place the device appropriately. Treatment will be administered for 1 hour per day for 4 weeks.
  Interventions: Device: High Frequency Impulse Therapy
- Sham arm (Sham Comparator): The sham unit looks identical to the experimental unit. There may be a sensation experienced by subjects with the sham device but it does not deliver an electric current as the experimental units. The study coordinator will assist each subject to place the device appropriately. Treatment will be administered for 1 hour per day for 4 weeks.
  Interventions: Device: High Frequency Impulse Therapy - Sham

INTERVENTIONS:
Device: High Frequency Impulse Therapy — The home TENS unit device is an at-home transcutaneous electrical nerve stimulation unit in that it provides non-invasive transcutaneous electrical impulses to reduce pain. It is a small, wearable device that utilizes both high and low frequencies to create a nerve-block effect based on the same gating theory.
  Other Names: Transcutaneous electrical nerve stimulation
  Arms: Experimental arm
Device: High Frequency Impulse Therapy - Sham — This device looks like the experimental device but does not provide the electrical current.
  Other Names: Transcutaneous electrical nerve stimulation - Sham
  Arms: Sham arm

SUMMARY:
The aim of this study is to determine whether self-administered, at-home use of a transcutaneous electrical nerve stimulating device is an effective, acceptable and feasible method of relief from neuropathic pain among patients with Neuromyelitis optica spectrum disorder (NMOSD).

DETAILED DESCRIPTION:
Neuromyelitis optica spectrum disorder (NMOSD) is a chronic relapsing autoimmune disease of the central nervous system (CNS) that preferentially targets the optic nerves and spinal cord, leading to paralysis, blindness and death. NMOSD is a rare disease that affects approximately 4,000-8,000 (8,000 - 15,000) people in the United States, disproportionately affects non-Caucasians and females, and has a worldwide prevalence estimated to be 0.52 to 4.4/100,000. Pain is a severely disabling component of the disease with up to 91% of patients reporting central neuropathic pain (CNP) characterized by agonizing burning, shooting or tingling sensation in the face, arms, torso and legs. NMOSD lesions in the spinal cord are characteristically long and destructive, and pain is more prevalent in NMOSD than in most other neurological diseases. Research on the impact of persistent pain on quality of life (QoL) in NMOSD has found that those patients with CNP experience more depression, less enjoyment of life, and more difficulty with ambulation. Currently, there is no standard of care for CNP treatment and off-label use of medications typically used for diabetic peripheral neuropathy are often insufficient. NMOSD is a devastating disease and there remains a high unmet need for effective treatment of CNP.

Transcutaneous electrical nerve stimulation (TENS) therapy is a non-invasive pain modifying intervention that utilizes transcutaneous electrical stimulation of ascending (sensory) fibers with the intent of re-organizing maladaptive signaling pathways. This neuromodulatory therapy has been investigated for treatment of persistent peripheral neuropathic pain in several conditions including chemotherapy-induced neuropathy, post-herpetic neuralgia and post-surgical neuropathic pain with promising results. Patients report sustained relief after undergoing daily treatment sessions for 10 consecutive weekdays.

Recently the investigators completed a sham controlled trial using a TENS unit called Scrambler in NMOSD patients showing a meaningful reduction in neuropathic pain compared to controls. The Scrambler device must be operated in an office by a professional technician, thereby limiting its usefulness to the wider NMOSD population. The home TENS device is similar to the Scrambler unit in that it provides non-invasive transcutaneous electrical impulses to reduce pain. It is a small, wearable device that utilizes both high and low frequencies to create a nerve-block effect based on the same gating theory. Because the TENS device for this study is programmable remotely, a controlled trial can be conducted while keeping the patient blinded to the trial arm.

For patients with NMOSD and other conditions that cause pain originating in the central nervous system, non-obtrusive, non-pharmacological devices might prove a viable alternative to pain medications. Pharmaceutical treatments for pain such as opioids have led to addiction and life-style changes with unacceptable side effects. Cost and side effects are concerns with other pharmacologic therapies for pain. In addition, in efforts to control pain, many patients are prescribed multiple medications, and then have to cope with the complexities and hazards of polypharmacy. Most importantly, none of the pharmaceutical treatments for pain in NMOSD have been proven effective in a trial.

If it can be shown among a significant patient cohort that a safe and effective at-home nonpharmacological pain therapy is available for patients with NMOSD, it would be life altering for a great many - not only those with NMOSD, but also with related neuroimmune disorders and other conditions with central neuropathic pain.

The goal of this project is to provide an effective, non-invasive treatment for neuropathic pain in NMOSD that can be safely employed at home. Many NMOSD patients have such chronic pain and/or disability that frequent visits to the clinic for therapy is difficult, if not impossible, in the best of times. Secondly, safe at-home treatments that offer continuous relief of pain (and potentially other co-occurring symptoms) can improve quality of life immensely during this, and likely future times of social distancing, when leaving home is dangerous, especially for a population on lifelong immune suppressants. Also, an at-home therapeutic option will save both time and money for patients.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18 years of age or older diagnosed with NMOSD per the 2015 NMOSD criteria
2. Patients must be positive for the aquaporin-4 antibody in serum.
3. Presence of persistent neuropathic pain (>3 months) rated at a level of 4 or higher on the Wong-Baker Faces Pain Scale
4. Patients must be stable in their disease, such that they have had no spinal cord relapses within 6 months prior to enrollment
5. Patients must be on a stable medication regimen that may include anti-epileptic, antidepressant, or non-steroidal anti-inflammatory medications, with no adjustments to the regimen within 30 days of enrollment
6. Pain must be localized to a spinal cord lesion
7. Patient understands the study regimen, its requirements, risks, and discomforts, and is able and willing to sign an informed consent form

Exclusion Criteria:

1. Patients who are cognitively or mentally incompetent
2. Any of the following: pregnant women, nursing women, women of childbearing potential or their sexual partners who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, abstinence, etc.).
3. Use of an investigational agent for pain control concurrently or within the past 30 days
4. History of an allergic reaction or previous intolerance to transcutaneous electronic nerve stimulation or to latex
5. Patients with implantable drug delivery systems, e.g. Medtronic Synchromed.
6. Patients with heart stents or metal implants such as pacemakers, automatic defibrillators, cochlear implants, aneurysm clips, vena cava clips and skull plates (Metal implants for orthopedic repair, e.g. pins, clips, plates, cages, joint replacements are allowed)
7. Patients with a known history of myocardial infarction or ischemic heart disease within the past six months
8. Prior celiac plexus block, or other neurolytic pain control treatment, within 1 month
9. Other identified causes of painful parasthesias existing prior to chemotherapy (e.g., carpal tunnel syndrome, B12 deficiency, AIDS, monoclonal gammopathy, diabetes, heavy metal poisoning amyloidosis, syphilis, hyperthyroidism or hypothyroidism, inherited neuropathy, etc.) that might be responsible for the patient's current neuropathic symptoms
10. Skin conditions such as open sores that would prevent proper application of the electrodes
11. Patients with an ongoing concomitant central neurologic disorder or history of epilepsy, brain damage, or symptomatic brain metastases
12. Other medical or other condition(s) that in the opinion of the investigators might compromise the objectives of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2025-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Levy, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vishnevetsky A, Romanow G, Levy M. A transcutaneous electrical nerve stimulation device for the relief of neuropathic pain in NMOSD: A randomized, double-blind, sham-controlled trial. Mult Scler J Exp Transl Clin. 2024 Dec 5;10(4):20552173241301018. doi: 10.1177/20552173241301018. eCollection 2024 Oct-Dec. PMID 39651334

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via social media outreach and directly in the clinic at the Neuroimmunology Clinic and Research Laboratory at Massachusetts General Hospital. The trial was entirely virtual, and the research coordinator screened potential participants by phone.
Pre-assignment Details: Inclusion criteria included age 18+ years, diagnosis of NMOSD, presence of aquaporin-4 immunoglobulin (AQP4 IgG) serum antibodies, pain lasting ≥ 3 months attributable to a previous inflammatory spinal cord lesion, and pain rated at a level of ≥ 4 on an 11-point Numeric Rating Scale (NRS).12 Exclusion criteria included spinal cord relapses or surgery to treat a pain-related condition within 6 months of enrollment, presence of neuropathic pain due to non-NMOSD-related identified causes.
Period: Overall Study
Arm/Group | Experimental Arm | Sham Arm
Started | 23 | 23
Completed | 19 | 21
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Population: There is no difference.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Arm | Sham Arm | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.6 (15.3) | 51.1 (13.2) | 52.4 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 19 | 19 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Score on the Numerical Rating Score (NRS)
Description: The NRS scale is an 11 point scale (0-10) with 0 as no pain and 10 as worst pain to determine the pain level. The result posted here is difference between the NRS at baseline and the NRS at 4 weeks.
Time Frame: 4 weeks from baseline to completion of the experimental phase.
Population: All individuals who completed their baseline and week 4 assessment were included in the analysis as randomized, regardless of actual device usage or further participation in the trial. Twenty-one participants in the sham arm and 19 in the TENS arm met these criteria.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Arm | Sham Arm
Number analyzed (Participants) | 19 | 21
units on a scale | 2.2 (2.2) | 1.3 (2.3)

2. Secondary Outcome: "Worst" Pain Score on the NRS Scale
Description: The NRS scale is an 11 point scale (0-10) with 0 as no pain and 10 as worst pain to determine the pain level. The result posted here is difference between the worst NRS at baseline and the worst NRS at 4 weeks.
Time Frame: 4 weeks from baseline to completion of the experimental phase.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Arm | Sham Arm
Number analyzed (Participants) | 19 | 21
units on a scale | 1.0 (2.1) | 1.4 (2.0)

3. Secondary Outcome: Withdrawal From Trial
Description: The number of patients who withdraw because of poor compliance.
Time Frame: 4 weeks from baseline to completion of the experimental phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm | Sham Arm
Number analyzed (Participants) | 23 | 23
Participants | 4 | 2

4. Secondary Outcome: Quality of Life Survey
Description: SF36 quality of life questionnaire summary score. The SF-36 scale range is from 0 to 100, with higher scores indicating better health and lower scores indicating poorer health across all eight domains measured by the survey; essentially, a score of 0 represents the worst possible health and 100 represents the best possible health.
Time Frame: 4 weeks from baseline to completion of the experimental phase.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Arm | Sham Arm
Number analyzed (Participants) | 19 | 21
score on a scale | 14.7 (13.5) | 10.2 (14.5)

ADVERSE EVENTS:
Time Frame: 2 years
Description: Addressing this issue: "The arms/groups appear inconsistent with information in other parts of the record. Each arm/group should be described separately, or a valid explanation provided."
  No adverse event data from the planned open label arm was collected. There is no data to report.
Arm/Group | Experimental Arm | Sham Arm
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 16/23 | 14/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Arm (N=23) | Sham Arm (N=23)
Increased pain (Nervous system disorders) | 3 | 4
Worsened vision (Nervous system disorders) | 1 | 0
Itchiness (Nervous system disorders) | 0 | 1
Insomnia (Nervous system disorders) | 0 | 1
Burning discomfort (Nervous system disorders) | 0 | 1
Restless Legs Syndrome (Nervous system disorders) | 0 | 1
Muscle twitching (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 1 | 1
Numbness (Nervous system disorders) | 1 | 1
Muscle spasms (Nervous system disorders) | 2 | 0
Phantom feelings (Nervous system disorders) | 3 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 3 | 2
Palpitations (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT04614454/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-14): https://cdn.clinicaltrials.gov/large-docs/54/NCT04614454/ICF_001.pdf